CLINICAL TRIAL: NCT03401710
Title: Erythropoietin Role in Acute Kidney Injury (EAKI): a Pragmatic Clinical Trial
Brief Title: Erythropoietin Role in Acute Kidney Injury
Acronym: EAKI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For very slow recruitment
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Mabel Aoun, MD, instructor, nephrology department, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAKI2017
Record Dates: First submitted 2017-12-06; First posted 2018-01-17 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Anemia Renal
Keywords: Anemia, Acute Kidney injury, ESA, Erythropoietin
MeSH Terms: conditions — Anemia; Acute Kidney Injury | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Recombinant human erythropoietin 4000 UI will be administered subcutaneously every other day
  Interventions: Drug: Erythropoietin
- Group 2 (No Intervention): No recombinant human erythropoietin will be administered to this group

INTERVENTIONS:
Drug: Erythropoietin — Erythropoietin 4000 UI will be administered every other day subcutaneously
  Other Names: No treatment
  Arms: Group 1

SUMMARY:
The use of erythropoietin to treat anemia in acute kidney injury (AKI) is controversial. No previous clinical trial has assessed the possible reduction of transfusions when erythropoietin is started very early in a setting of in-hospital acute kidney injury.

This randomised multicenter pragmatic clinical trial will compare the need for transfusion in acute kidney injury between two groups: group 1 will receive erythopoietin 4000 UI every other day and group 2 the usual treatment.

DETAILED DESCRIPTION:
Introduction

Background and rationale

Since the release of the recombinant human erythropoietin (rhuEPO) at the beginning of the 90s, transfusions are less needed to treat anemia in chronic kidney disease patients. This has been a major revolution in the management of renal anemia in chronic kidney disease and led to a tremendous decrease in hepatitis B and C transmissions in dialysis patients.

However the use of rHuEPO to treat anemia in acute kidney injury (AKI) is controversial. AKI is a common disease with a worldwide incidence estimated at 21% and a trend to be higher in the critical care setting.

The Kidney Disease Improving Global Outcomes (KDIGO) work group combined the RIFLE and AKIN classifications of AKI. Therefore, AKI has been defined as an increase in serum creatinine (SCr) ≥0.3 mg/dL (≥26.5 μmol/L) within 48 h or an increase in SCr to ≥1.5 times baseline within the last 7 days or a urine volume of <0.5 mL/kg/h for 6 hours.

As it was already shown, the majority of patients admitted with AKI have anemia (91% in Hales et al study) and the anemia seems to be related to the degree of oliguria and uremia level. Erythropoietin is secreted at the tubulo-interstitial level and it has been shown that a chronic injury would lead to a decrease in erythropoietin secretion. Some studies have shown that erythropoietin level increases the first 48 hours of acute kidney injury then decreases progressively. Transfusions are needed when critically ill patients stay at the hospital for a long period of time. And transfusions during acute kidney injury may lead to sensitization and cause limitation for future transplantation in patients who reach end-stage renal disease. Therefore prevention of transfusions in acute kidney injury patients is highly needed.

A search of the literature for "human recombinant erythropoietin" and "acute renal failure" or "acute kidney disease" or "acute kidney injury" did not reveal any clinical trial or observational study targeting this issue. Some studies assessed the role of rHuEPO to prevent acute kidney injury in cardiac surgery patients and contrast-induced nephropathy with conflicting results. Some experimental studies on rats demonstrated a favorable effect of rHuEPO and darbepoetin on the ischemic renal injury. A recent metaanalysis of 10 randomized controlled trials showed no beneficial effect of erythropoietin on preventing AKI or dialysis or death but the majority of patients received a single dose of rHuEPO.

The role of rHuEPO after the occurrence of acute kidney injury is not well studied. One retrospective study in 2005 showed that rHuEPO administration in acute renal failure patients did not decrease the transfusion requirements. However it included many limitations such as the low dose of rHuEPO used, the absence of preset hemoglobin level threshold for blood transfusions. A recent clinical trial in children with hemolytic uremic syndrome showed a decrease in transfusion in patients receiving EPO. Therefore a clinical trial taking into account all of these factors would be more conclusive regarding the exact role of erythropoietin in acute kidney injury patients.

Trial objectives The primary objective of this trial is to compare the number of red blood cell transfusions in patients with acute kidney injury and anemia whether receiving or not rHuEPO.

The secondary objectives are a) to compare the renal survival between the two groups, b) to compare the patient survival between the two groups.

Trial design This is a randomized, controlled, multicenter, pragmatic clinical trial. Patients will be randomized to one of two arms and then group one will receive the rHuEPO and group two the usual treatment.

This study will assess the superiority of rHuEPO use in acute kidney injury with anemia against no use of rHuEPO.

Methods: Data collection, management, and analysis

Data collection methods Data collection will be carried out using excel program. Data for presumed cause of acute kidney injury, comorbidities, medications and laboratory results are collected from the patients' medical records. The following variables will be studied: age, gender, body mass index (BMI), diabetes, smoking in the last year, hypertension, hyperlipidemia, previous cardiovascular disease, previous inflammatory disease, previous chronic obstructive pulmonary disease (COPD), previous serum creatinine (Scr) and Scr on admission (with corresponding eGFR using the CKD-EPI equation), phosphate, calcium, albumin, bicarbonate, hemoglobin, ferritin, TSAT, vitamin B12, uric acid and CPK. Data on previous medications will be collected: iron substitutes, multivitamins, non-steroidal anti-inflammatory drugs, antihypertensive medications such as ACE inhibitors and ARBs, antiplatelet agents, urate lowering therapy, antibiotics and corticosteroids.

Definitions Acute kidney injury is defined based on the RIFLE, AKIN and KDIGO criteria. Anemia is defined in general as Hb <13 g/dl in male patients and <12 g/dl in females. Anemia in this trial will be defined as Hb<11 g/dl.

Coronary artery disease is defined as a history of myocardial infarction or obstructive coronary artery disease, treated medically or interventionally. Diabetes and hypertension are defined as taking antidiabetic treatment or antihypertensive treatment respectively.

Statistical analysis Continuous variables will be presented as mean ± standard deviation (SD). Differences between the study groups will be tested using χ2 tests (for categorical variables). Bivariate correlation analysis will be performed using the Pearson's correlation coefficient. The Kaplan-Meier method will be used to estimate the cumulative survival. Cox regression will be used to determine the effect of erythropoietin on renal survival and total mortality. Statistical analysis will be performed with SPSS. A P-value of ≤0.05 is considered statistically significant.

Methods: Monitoring

Data monitoring Follow-up with laboratory measurements and medication dosage Hemoglobin and creatinine will be measured with the standard laboratory techniques every day. C-reactive protein (CRP) will be measured at least twice.

Medications administered during the hospitalization will be collected as the total dose of the duration of stay, particularly noradrenaline, dopamine, furosemide, antibiotics, anticoagulants, vitamins, enteral or parenteral nutrition, proton-pump inhibitors.

Transfusions: quantity of units of packed red blood cells, platelets, fresh frozen plasma will be collected.

Clinical follow-up Data including daily systolic and diastolic blood pressure, average hospital length of stay (LOS), oligo-anuria at any stage of the AKI, need for dialysis and number of days till serum creatinine starts to decrease will be collected.

Adverse events will be also reported such as any thrombotic event.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years old hospitalized with acute kidney injury and anemia

Exclusion Criteria:

* pregnant women, terminally ill patients, patients with major or minor thalassemia, patients with stable chronic kidney disease or patients on dialysis and patients who were receiving rHuEPO or any erythropoiesis-stimulating agent (ESA) before admission.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Transfusion | Admission- One month
  Number of red blood cell transfusions

SECONDARY OUTCOMES:
Renal survival | Admission - One month
  Creatinine level at discharge
Mortality | Admission - One month
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Mabel Aoun, MD, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint Georges Hospital, Ajaltoun, Ajaltoun, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aoun M, Sleilaty G, Boueri C, Younes E, Gabriel K, Kahwaji RM, Hilal N, Hawi J, Araman R, Chelala D, Beaini C. Erythropoietin in Acute Kidney Injury (EAKI): a pragmatic randomized clinical trial. BMC Nephrol. 2022 Mar 13;23(1):100. doi: 10.1186/s12882-022-02727-5. PMID 35279078